CLINICAL TRIAL: NCT04780217
Title: A Phase 1/2a Open-Label Dose Escalation and Dose Expansion Study of T3011 When Administered Intravenously as a Single Agent and in Combination With Other Therapy in Subjects With Advanced Solid Tumors
Brief Title: Intravenous T3011 Given as a Single Agent and in Combination With Other Therapy in Subjects With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ImmVira Pharma Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MVR-T3011-003
Record Dates: First submitted 2021-02-06; First posted 2021-03-03 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Solid Tumor; Hepatocellular Carcinoma; Colorectal Cancer; NSCLC; Ovarian Cancer; Endometrial Cancer
Keywords: solid tumor
MeSH Terms: conditions — Carcinoma, Hepatocellular; Colorectal Neoplasms; Ovarian Neoplasms; Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phase 1 (Experimental): T3011 Single Agent Dose Escalation in participants with solid tumors
  Interventions: Biological: T3011

INTERVENTIONS:
Biological: T3011 — T3011 will be administered through IV drip or pumping.

SUMMARY:
A Phase 1/2a Open-Label Dose Escalation and Dose Expansion Study of T3011 when Administered Intravenously as a Single Agent and in Combination with Other Therapy in Subjects with Advanced Solid Tumors

DETAILED DESCRIPTION:
This is a multicenter, open-label study conducted in two phases (as outlined in the subsections below):

Phase 1: T3011 administered intravenously as a single agent in subjects with pathologically confirmed locally recurrent or metastatic solid tumors, who have failed or declined SOC treatment. Phase 1 will use a 3+3 design to evaluate escalating doses of single agent T3011. Cohorts of three subjects will be enrolled at each T3011 dose level with expansion to six subjects, if necessary, to assess toxicity. Total enrollment will depend on the toxicities observed, with approximately 36-42 evaluable subjects enrolled in phase 1.

Phase 2a: An expansion study will be conducted based on phase 1 results.

ELIGIBILITY:
Inclusion Criteria:

All subjects must meet the following criteria for inclusion:

1. Subjects with one of the following cancers:

   • Pathologically confirmed, locally recurrent or metastatic solid tumors, including, but not limited to NSCLC, hepatocellular carcinoma, colorectal cancer, ovarian cancer and endometrial cancer (Phase 1).
2. Disease progression on or unlikely to respond to SOC therapy at the discretion of the Investigator. SOC may include, but is not limited to, chemotherapy, targeted therapy or immunotherapy.
3. Age 18 years or older.
4. At least one target lesion per RECIST version 1.1.

   • A previously irradiated lesions can be considered as target lesion only if PD has been unequivocally documented at that site since radiation.
5. Eastern Cooperative Oncology Group (ECOG) performance status 0 - 1.
6. Life expectancy ≥ 12 weeks.
7. Adequate bone marrow function defined by absolute neutrophil count (ANC) of ≥ 1.5 × 109/L, platelet count of ≥ 100 × 109/L, and hemoglobin (Hb) of ≥ 8.5 g/dL.
8. Adequate hepatic function defined as aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 3 × upper limit of normal (ULN) and total bilirubin ≤ 1.5 × ULN (except subjects with Gilbert's Syndrome, wherein total bilirubin < 3.0 mg/dL is acceptable).
9. Adequate renal function defined as creatinine clearance > 50 mL/min as determined by the Cockcroft-Gault equation.
10. Female subjects must be surgically sterile (or have a monogamous partner who is surgically sterile), or be at least 2 years postmenopausal, or commit to using 2 acceptable forms of birth control (defined as the use of an intrauterine device, a barrier method with spermicide, condoms, any form of hormonal contraceptives, or abstinence) for the duration of the study and for 6 months following the last dose of study treatment. Male subjects must be sterile (biologically or surgically) or commit to the use of a reliable method of birth control (condoms with spermicide) for the duration of the study and for 6 months following the last dose of study treatment.
11. Women of childbearing potential (WCBP) must have a negative serum pregnancy test at Screening within 14 days of dosing with T3011 and a negative urine pregnancy test pre-dose on C1D1 (assessment not required at C1D1 if completed within the previous 7 days of C1D1).

    Note: A woman is considered to be of childbearing potential if she is postmenarchal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and is not permanently infertile due to surgery (i.e., removal of ovaries, fallopian tubes, and/or uterus) or another cause as determined by the investigator (e.g., Müllerian agenesis).
12. Last dose of previous anticancer therapy ≥ 21 days; radiotherapy > 14 days (except prior focal palliative radiotherapy must have been completed at least 1 week prior to the first dose of study treatment); major surgery > 21 days; or last dose of therapy with tyrosine kinase inhibitors within 5 times the half-life of the inhibitor prior to first dose of study treatment. Last dose of checkpoint inhibitor ≥ 14 days, as long as treatment related toxicities resolve to ≤ Grade 1.
13. Resolution of all prior anticancer therapy toxicities (except for alopecia) to ≤ CTCAE version 5.0 Grade 1.

    Note: subjects with immune-mediated endocrinopathies on replacement therapy are eligible. Subjects with toxicities attributed to the prior anticancer therapy and not expected to resolve, such as neuropathy or ototoxicity after platinum-based therapy, are permitted to enroll. Subjects with other toxicities > CTCAE version 5.0 Grade 1 may be enrolled with approval from the sponsor.
14. Willingness to provide pre- and post-treatment fresh tumor biopsy specimens, if tumor is easily accessible, as specified in the Schedule of Assessments. Subject is eligible to participate without providing fresh tumor biopsy specimens, with approval from the Medical Monitor.
15. Capable of understanding and complying with protocol requirements.
16. Signed and dated institutional review board/independent ethics committee (IRB/IEC) approved informed consent form (ICF) before any protocol-directed screening procedures are performed.

Exclusion Criteria:

Subjects are to be excluded from the study if they meet any of the following criteria:

1. Prior treatment with another OV (including T-VEC), tumor vaccines, cellular therapy or gene therapy.
2. Prior treatment with anti-PD-(L)1 monoclonal antibody in combination with IL-12.
3. Subjects with rapidly disease progression, defined as subjects who cannot tolerate interruption of systemic antitumor therapy for at least 8 weeks, according to the investigator's judgment.
4. Previous intolerance to anti-PD-(L)1 monoclonal antibody or previous history of immunotherapy induced non-infectious pneumonitis/interstitial lung disease.
5. Requires continued concurrent systemic therapy with any drug active against HSV (acyclovir, valaciclovir, penciclovir, famciclovir, ganciclovir, foscarnet, cidofovir). Topical use of drugs against HSV are allowed.
6. Live, attenuated vaccines within 4 weeks prior to initiation of study treatment (subjects vaccinated with inactivated vaccines can be enrolled).
7. Primary or acquired immunodeficient states (leukemia, lymphoma, human immunodeficiency virus [HIV]/acquired immunodeficiency syndrome [AIDS]).
8. Active infection requiring systemic treatment.
9. Pregnant or lactating.
10. Splenectomy, previous allogenic tissue/solid organ transplant.
11. Positive serological test of hepatitis B virus (HBV) or hepatitis C virus at Screening.

    * Subjects who test positive for anti-hepatitis C antibody (anti-HCV) but negative for HCV ribonucleic acid (RNA) are considered eligible to participate in the study.
    * Subjects with infection of hepatitis B (positive hepatitis B surface antigen [HBsAg] result) will be excluded. Subjects with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [HBcAb] and absence of HBsAg) are eligible.
12. Active autoimmune disease or other medical conditions (e.g., active interstitial lung disease/pneumonitis or eczema, psoriasis, or other clinically significant dermatologic disorders) requiring chronic systemic steroid (> 10 mg/day prednisone or equivalent) or immunosuppressive therapy within 4 weeks prior to first administration of study treatment (unless agreed otherwise between the Medical Monitor and the Investigator on a case-by-case basis). Non-systemic corticosteroids (eg, topical, inhaled) are allowed.
13. Subjects with untreated and/or symptomatic metastatic central nervous system (CNS) disease, primary CNS tumors, leptomeningeal disease or spinal cord compression. However, subjects with brain/CNS metastases who have undergone surgery or radiotherapy, whose disease is stable and who have been on a stable dose of corticosteroids (≤ 10 mg prednisone or equivalent) for at least 4 weeks prior to the first administration of study treatment will be eligible.
14. History of another primary malignant tumor, except the following: 1) the patient has undergone potentially curative therapy with no evidence of that disease and recurrence for 3 years prior to the first dose of study treatment; 2) Adequately treated non-melanoma skin cancer or lentigo with no evidence of malignancy; 3) Adequately treated carcinoma in situ without evidence of disease.
15. Subjects with moderate to large amount of pleural effusion, ascites or pericardial effusion who need drug or medical intervention. Subject may be eligible to participate following discussion with investigator and approval from the sponsor.
16. Unexplained >38.5℃ fever (If the fever is caused by the tumor according to the investigator's judgment, the patient can be enrolled) occurs during the screening period or on the day of administration, which in the judgment of investigator, would interfere with patient participation in the study or evaluation of patient's efficacy.
17. History of seizure disorders within 6 months prior to Screening.
18. Active oral or skin herpes lesion at Screening.
19. Plan to receive any other anti-tumor therapy (including herbal therapy that has anti-tumor effects) during treatment with study drug.
20. History of congestive heart failure (> New York Heart Association Class II), active coronary artery disease, unevaluated new onset angina within 3 months or unstable angina (angina symptoms at rest), or clinically significant cardiac arrhythmias.
21. History of allergic reactions attributed to compounds of similar biological composition to HSV-1, IL-12, or anti-PD-1 monoclonal antibody or their excipients.
22. History of psychiatric disorders that would interfere with cooperation with the requirements of the trial or is still requiring for medication control.
23. History of substance abuse (including alcohol) within 6 months prior to signing informed consent.
24. Other systemic conditions or organ abnormalities that, in the opinion of the Investigator, may interfere with the conduct and/or interpretation of the current study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-08-10 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of escalating doses of single agent IV T3011 Characterize DLTs and identify the MTD and/or the RP2D of single agent IV T3011 | Up to 2 years from first dose of T3011
  Number of participants with Adverse Events (TEAEs, SAEs, AESIs), with abnormal clinically significant vital signs, with abnormal physical examination findings and abnormal laboratory tests results

SECONDARY OUTCOMES:
Evaluate the immunogenicity of single agent IV T3011. | Up to 2 years from first dose of T3011
  Measurement of ADAs and Nabs of IL-12, anti-PD-1 antibody and HSV-1 (test Nabs when ADAs are positive).
Overall response rate (ORR) | Up to 2 years from first dose of T3011
  Defined as the percentage of subjects who have best overall response (BOR) as CR or partial response (PR), as determined according to RECIST v1.1. CR or PR will be claimed only if the criteria for each are met at a subsequent time point at 4-8 weeks later.
Disease control rate (DCR) | Up to 2 years from first dose of T3011
  Defined as the percentage of subjects who have BOR as CR or PR or stable disease (SD) (if a subject develops SD, it needs to be confirmed at least 6 weeks later, that is, SD lasts at least 6 weeks), as determined according to RECIST v1.1.
Duration of response (DOR) | Up to 2 years from first dose of T3011
  Defined as the time from the first occurrence of a documented objective response to disease progression or death from any cause (whichever comes first), as determined according to RECIST v1.1
Progression-free survival (PFS) | Up to 2 years from first dose of T3011
  Defined as the time from the date of first treatment to the first occurrence of disease progression or death from any cause (whichever comes first), as determined according to RECIST v1.1.
Overall Survival (OS) | Up to 2 years from first dose of T3011
  OS is defined as the time from enrollment to death from any cause.
time to treatment failure（TTF） | Up to 2 years from first dose of T3011
  Defined as a composite endpoint measuring time from the date of first treatment to discontinuation of treatment for any reason, including disease progression, treatment toxicity, and death.
PFS2 | Up to 2 years from first dose of T3011
  Defined as the time from the date of initiation of new antitumor therapy to the first occurrence of disease progression after new antitumor therapy or death from any cause (whichever comes first)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Banner MD Anderson Cancer Center, Phoenix, Arizona
  - BRCR Medical Center Inc, Plantation, Florida
  - Prisma Health - Upstate, Greenville, South Carolina
  - Virginia Cancer Specialists, Greenville, South Carolina
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Mary Crowley Cancer Research, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: ImmVira Pharma Co. LTD — https://immviragroup.com/